CLINICAL TRIAL: NCT03563846
Title: Prospective, Open-Label, Randomized, Two-Period, Two-Sequence, Crossover Study Comparing RP-G28 Administered in the Fasted State and the Effect of a Standard Meal on the Pharmacokinetic Profile of RP-G28 in Healthy Volunteers
Brief Title: Effect of a Standard Meal on the Pharmacokinetic Profile of RP-G28 in Healthy Adult Male and Female Subjects
Acronym: RP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ritter Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G28-005
Record Dates: First submitted 2018-04-02; First posted 2018-06-20 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-06

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — RP-G28

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RP-G28 administered in the fasted state (Experimental): RP-G28, 15 g dissolved in water, administered in the fasted state
  Interventions: Drug: RP-G28
- RP-G28 administered in the fed state (Experimental): RP-G28, 15 g dissolved in water, administered immediately following the consumption of a standard non-dairy meal
  Interventions: Drug: RP-G28

INTERVENTIONS:
Drug: RP-G28 — RP-G28 is a purified galacto-oligosaccharide (GOS) product
  Other Names: galactic-oligosaccharide

SUMMARY:
Randomized, open-label, 2-period, 2-sequence, crossover study to evaluate the effect of a standard meal on the pharmacokinetic (PK) profile of orally administered RP-G28.

DETAILED DESCRIPTION:
This randomized, open-label, 2-period, 2-sequence, crossover study is designed to evaluate the effect of a standard meal on the pharmacokinetic (PK) profile of orally administered RP-G28, which is being developed for the treatment of lactose intolerance. The study consists of a screening visit (during the interval from Day -21 to Day -3), baseline/check-in to the clinical research unit (Day -2 to Day -1), 2 treatment periods (Day 1 and Day 3), a 48-hour washout between doses, check-out from the clinical research unit (Day 4), and 1 follow-up phone call conducted 7 to 10 days after the final dose of the study drug (i.e., during the interval from Day 10 to Day 13). The duration of subject study participation is approximately 5 weeks. Plasma samples for PK analysis will be taken at specified timepoints from 24 hours prior to each dose through 24 hours after each dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects between 18 and 60 years of age
2. Subjects with body weights greater than or equal to 50 kg and a body mass index (BMI) between 18 kg/m2 and 32 kg/m2
3. Female subjects of childbearing potential and males and their female partner(s) of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 30 days after the end of the study

Exclusion Criteria:

1. Pregnant or lactating females or male partners of females who are pregnant or lactating.
2. Subjects with any history of clinically significant bronchopulmonary, cardiovascular, cerebrovascular, hematologic, renal, hepatic, neurological, psychiatric, metabolic, or endocrine (eg, diabetes or thyroid disease) disease/disorder.
3. Use of prescription or over-the-counter (OTC) drugs, including vitamins and herbal or dietary supplements within 2 weeks (4 weeks for enzyme inducers including St. John's Wort) or 5 half-lives (whichever is longer), prior to the baseline/check-in visit, unless in the opinion of the investigator, prior use of the medication will not interfere with the study procedures or compromise subject safety.
4. Subjects with sustained supine or semi-supine systolic blood pressure of < 90 or > 140 mm Hg and supine or semi-supine diastolic blood pressure of < 50 or > 90 mm Hg at the screening or baseline/check-in visits.
5. Subjects with a resting heart rate of < 45 or > 100 beats per minute at the screening or baseline/check in visits.
6. Subjects with any clinically relevant deviation from normal during the physical examination, including vital signs at the screening or baseline/check-in visits.
7. Subjects with a known history of hypercalcemia, hyperparathyroidism, or hypervitaminosis D.
8. Use of calcium or vitamin D supplements (prescription or OTC) within 2 weeks prior to the baseline/check-in visit.
9. Subjects with a history of allergic reactions or hypersensitivities to galacto-oligosaccharides or any significant drug-related or food-related allergy (such as anaphylaxis or hepatotoxicity).
10. Regular use of probiotics, antacids, histamine type 2 (H2)-receptor blockers, proton pump inhibitors, or any medications that may alter the normal gastric environment and/or motility, or use of such medications within 2 weeks prior to the baseline/check-in visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 extrapolated to infinity | Days 2 and 1 pretreatment; Day 1 post-treatment, Day 1-3 washout, Day 3 and 4 post-treatment
  Assess systemic exposure of RP-G28 when administered in the fed and fasted state

SECONDARY OUTCOMES:
Adverse events | 2, 3, 2 and 1 days pretreatment; 1 - 13 days post-treatment
  Adverse events will be continuously monitored throughout the entire study, including follow-up.
Serum chemistry | 21 and 3 days pretreatment; day 4 post-treatment
  Albumin, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, blood urea nitrogen, calcium, chloride, carbon dioxide, creatinine, total bilirubin, gamma glutamyl transferase, glucose, lactic dehydrogenase (lactate dehydrogenase), phosphorus, potassium, sodium, total cholesterol, total protein, uric acid, and vitamin D.
Hematology | 21 and 3 days pretreatment; day 4 post-treatment
  Number of subjects with abnormal laboratory values will be flagged and summarized separately
Urinalysis | 2, 3, 2 and 1 days pretreatment; day 1 and 3 post-treatment
  Number of subjects with abnormal laboratory values will be flagged and summarized separately

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Pearson, PhD, Study Director — Ritter Pharmaceuticals
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No